CLINICAL TRIAL: NCT00976703
Title: Weighted Bag Versus Inner Thigh Taping for Cervical Ripening With a Foley Catheter Prior to an Induction of Labor
Brief Title: Foley Bulb Traction for Cervical Ripening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Kelly S Gibson, Physician, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB09-00392
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-05

CONDITIONS: Cervical Ripening; Induction of Labor
Keywords: cervical foley catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- weighted bag (Active Comparator): For the weighted bag, a 500cc saline bag will be taped to an empty Foley bag which will be attached to the cervical Foley catheter. This bag will then be placed to gravity over the end of the bed. The bed will be raised so that the bag does not touch the floor. The foley and the bag will be re-assessed every 30min by the nursing staff.
  Interventions: Other: weighted bag
- leg taping (Active Comparator): For the leg taping, the cervical foley catheter will be pulled to gentle traction and attached to the patient's inner thigh using a reclosable foley catheter fastener. The foley catheter and the traction will be assessed every 30min by the nursing staff. The tension will be renewed and the Foley re-adjusted if necessary at each check.
  Interventions: Other: leg taping

INTERVENTIONS:
Other: weighted bag — For the weighted bag, a 500cc saline bag will be taped to an empty Foley bag which will be attached to the cervical Foley catheter. This bag will then be placed to gravity over the end of the bed. The bed will be raised so that the bag does not touch the floor. The foley and the bag will be re-assessed every 30min by the nursing staff.
  Arms: weighted bag
Other: leg taping — For the leg taping, the cervical foley catheter will be pulled to gentle traction and attached to the patient's inner thigh using a reclosable foley catheter fastener. The foley catheter and the traction will be assessed every 30min by the nursing staff. The tension will be renewed and the Foley re-adjusted if necessary at each check.
  Arms: leg taping

SUMMARY:
This study aims to determine what type of traction, weighted bag or inner thigh taping, on foley catheters for cervical ripening results in a greater cervical dilation and shorter length of labor.

The primary outcomes are post-ripening dilation of 3 cm or more and time to delivery.

The secondary outcomes are patient pain/comfort rating and method of delivery. The investigators hypothesize that the use a weighted bag will result in a 20% increase in post-ripening dilation of at least 3 cm and a shorter average length of labor.

DETAILED DESCRIPTION:
Over the last 20 years the number of induced labors doubled so that over one in five births in 2003 was induced. In response to the rising need for cervical ripening the American College Obstetricians and Gynecologists have stated that both mechanical and prostaglandin ripening is acceptable and safe.

Prior to beginning an induction, the Bishop score (cervical dilation, effacement, station, consistency, and position) is assessed. With Bishop scores less than five, a cervical ripening agent is commonly used. The mechanical dilation with a foley catheter works by both a direct stretching of the lower uterine segment and cervix and a local inflammatory response that releases matrix metalloproteinases and prostaglandins. It is often chosen due to its lower cost, low incidence of systemic side effects, and low risk of hyperstimulation.

Compared to misoprostol a foley with oxytocin was more effective at induction in primiparous patients, more effective at improving the dilation, safe to use after misoprostol, and not associated with an increased risk of uterine rupture in a vaginal birth after cesarean (VBAC). The foley was also shown to have a shorter induction time and less contractile abnormalities than prostaglandin E2 gel and no increased rate of uterine rupture in VBAC attempts. The use of extra-amniotic saline infusion with a foley catheter has been used to augment the mechanical stretching, however this did not decrease the induction time or improve the outcomes. Finally, a Cochrane Database review found that mechanical methods of cervical ripening were equally effective as prostaglandin agents.

Although the safety, efficacy, and side effects of foley catheter ripening have been compared with multiple other methods for cervical ripening, very few studies have compared different protocols for foley placement. One study showed that the use of oxytocin while the foley catheter was in place did not significantly shorten the time to delivery. Levy et al showed that a larger, 80 ml, balloon resulted in a greater post-ripening dilation and a higher number of deliveries in 24hours. No study to date has examined how the traction placed on the foley catheter affects the outcome.

Therefore, we propose doing a randomized controlled study in which the control is the current standard of care at MetroHealth Medical Center of placing a 500cc weight on the foley and placing it to gravity over the end of the bed. The comparison will be the method used at many institutions where the foley catheter is placed on gentle traction and taped to the inner thigh of the patient.

The primary outcomes measured will be a post-ripening dilation of 3cm or more and time to delivery. The secondary outcomes are patient pain/comfort rating and method of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Single viable intrauterine pregnancy
* Cephalic presentation
* Bishop score <6
* Need for induction of labor

Exclusion Criteria:

* Multiple gestation
* Bishop score >6
* Spontaneous labor/regular contractions on admission
* Rupture of membranes
* Previous uterine scar
* Grandmultiparity (greater than 5 deliveries)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Curtin SC, Park MM. Trends in the attendant, place, and timing of births, and in the use of obstetric interventions: United States, 1989-97. Natl Vital Stat Rep. 1999 Dec 2;47(27):1-12. PMID 10598437
- [Background] Martin JA, Hamilton BE, Sutton PD, Ventura SJ, Menacker F, Munson ML. Births: final data for 2003. Natl Vital Stat Rep. 2005 Sep 8;54(2):1-116. PMID 16176060
- [Background] Riskin-Mashiah S, Wilkins I. Cervical ripening. Obstet Gynecol Clin North Am. 1999 Jun;26(2):243-57. doi: 10.1016/s0889-8545(05)70072-3. PMID 10399759
- [Background] Gelber S, Sciscione A. Mechanical methods of cervical ripening and labor induction. Clin Obstet Gynecol. 2006 Sep;49(3):642-57. doi: 10.1097/00003081-200609000-00022. PMID 16885669
- [Background] Abramovici D, Goldwasser S, Mabie BC, Mercer BM, Goldwasser R, Sibai BM. A randomized comparison of oral misoprostol versus Foley catheter and oxytocin for induction of labor at term. Am J Obstet Gynecol. 1999 Nov;181(5 Pt 1):1108-12. doi: 10.1016/s0002-9378(99)70090-6. PMID 10561627
- [Background] Adeniji AO, Olayemi O, Odukogbe AA. Intravaginal misoprostol versus transcervical Foley catheter in pre-induction cervical ripening. Int J Gynaecol Obstet. 2006 Feb;92(2):130-2. doi: 10.1016/j.ijgo.2005.10.010. Epub 2005 Dec 2. No abstract available. PMID 16325816
- [Background] Caliskan E, Dilbaz S, Gelisen O, Dilbaz B, Ozturk N, Haberal A. Unsucessful labour induction in women with unfavourable cervical scores: predictors and management. Aust N Z J Obstet Gynaecol. 2004 Dec;44(6):562-7. doi: 10.1111/j.1479-828X.2004.00321.x. PMID 15598298
- [Background] Sciscione AC, Nguyen L, Manley J, Pollock M, Maas B, Colmorgen G. A randomized comparison of transcervical Foley catheter to intravaginal misoprostol for preinduction cervical ripening. Obstet Gynecol. 2001 Apr;97(4):603-7. doi: 10.1016/s0029-7844(00)01186-8. PMID 11275035
- [Background] Bujold E, Blackwell SC, Gauthier RJ. Cervical ripening with transcervical foley catheter and the risk of uterine rupture. Obstet Gynecol. 2004 Jan;103(1):18-23. doi: 10.1097/01.AOG.0000109148.23082.C1. PMID 14704239
- [Background] Sciscione AC, McCullough H, Manley JS, Shlossman PA, Pollock M, Colmorgen GH. A prospective, randomized comparison of Foley catheter insertion versus intracervical prostaglandin E2 gel for preinduction cervical ripening. Am J Obstet Gynecol. 1999 Jan;180(1 Pt 1):55-60. doi: 10.1016/s0002-9378(99)70149-3. PMID 9914578
- [Background] Ben-Aroya Z, Hallak M, Segal D, Friger M, Katz M, Mazor M. Ripening of the uterine cervix in a post-cesarean parturient: prostaglandin E2 versus Foley catheter. J Matern Fetal Neonatal Med. 2002 Jul;12(1):42-5. doi: 10.1080/jmf.12.1.42.45. PMID 12422908
- [Background] Lin MG, Reid KJ, Treaster MR, Nuthalapaty FS, Ramsey PS, Lu GC. Transcervical Foley catheter with and without extraamniotic saline infusion for labor induction: a randomized controlled trial. Obstet Gynecol. 2007 Sep;110(3):558-65. doi: 10.1097/01.AOG.0000278077.30890.87. PMID 17766600
- [Background] Guinn DA, Davies JK, Jones RO, Sullivan L, Wolf D. Labor induction in women with an unfavorable Bishop score: randomized controlled trial of intrauterine Foley catheter with concurrent oxytocin infusion versus Foley catheter with extra-amniotic saline infusion with concurrent oxytocin infusion. Am J Obstet Gynecol. 2004 Jul;191(1):225-9. doi: 10.1016/j.ajog.2003.12.039. PMID 15295370
- [Background] Boulvain M, Kelly A, Lohse C, Stan C, Irion O. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2001;(4):CD001233. doi: 10.1002/14651858.CD001233. PMID 11687101
- [Background] Pettker CM, Pocock SB, Smok DP, Lee SM, Devine PC. Transcervical Foley catheter with and without oxytocin for cervical ripening: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1320-6. doi: 10.1097/AOG.0b013e31817615a0. PMID 18515515
- [Background] Levy R, Kanengiser B, Furman B, Ben Arie A, Brown D, Hagay ZJ. A randomized trial comparing a 30-mL and an 80-mL Foley catheter balloon for preinduction cervical ripening. Am J Obstet Gynecol. 2004 Nov;191(5):1632-6. doi: 10.1016/j.ajog.2004.03.033. PMID 15547534
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Gibson KS, Mercer BM, Louis JM. Inner thigh taping vs traction for cervical ripening with a Foley catheter: a randomized controlled trial. Am J Obstet Gynecol. 2013 Sep;209(3):272.e1-7. doi: 10.1016/j.ajog.2013.05.028. Epub 2013 Jun 6. PMID 23685080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We performed a single-site randomized controlled trial at MetroHealth Medical Center, a tertiary hospital, from December 2009 to July 2012.
Pre-assignment Details: Eligibility criteria included: admission for an induction of labor, a fetus in cephalic presentation, and an unripe cervix defined as a Bishop score ≤ 6.
Groups:
- Weighted Bag (Traction): For the weighted bag, a 500cc saline bag will be taped to an empty Foley bag which will be attached to the cervical Foley catheter. This bag will then be placed to gravity over the end of the bed. The bed will be raised so that the bag does not touch the floor. The foley and the bag will be re-assessed every 30min by the nursing staff.
- Leg Taping (Taping): For the leg taping, the cervical foley catheter will be pulled to gentle traction and attached to the patient's inner thigh using a reclosable foley catheter fastener. The foley catheter and the traction will be assessed every 30min by the nursing staff. The tension will be renewed and the Foley re-adjusted if necessary at each check.
Period: Overall Study
Arm/Group | Weighted Bag (Traction) | Leg Taping (Taping)
Started | 99 | 98
Completed | 96 | 95
Not Completed | 3 | 3
Not completed — Physician Decision | 1 | 1
Not completed — ineligible for study | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weighted Bag (Traction) | Leg Taping (Taping) | Total
Number analyzed (Participants) | 99 | 98 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 97 | 96 | 193
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.7 (6.9) | 25.5 (5.9) | 25.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 98 | 197
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 99 | 98 | 197

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery
Time Frame: an average of 20 hours, up to 40 hours
Population: In order to find a 20% difference with a 40% standard deviation, power of 90%, and alpha of 0.05, we estimated we needed 86 patients in each arm. We aimed to recruit 194 patients to account for potential dropouts and missing data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Weighted Bag (Traction) | Leg Taping (Taping)
Number analyzed (Participants) | 96 | 95
hours | 19.8 (8.5) | 18.8 (8.0)

2. Secondary Outcome: Patient Pain/Comfort Rating
Description: Using a visual analog pain scale, with 0 being no pain and 10 being the most severe pain possible, the patients were asked to assess their pain every hour. The highest pain score recorded while the Foley catheter was in place was used. The data are reported as the median and range.
Time Frame: an average of 20 hours, up to 40 hours
Population: All patients had pain scores recorded and used in analysis. The values in the table represented the recorded data available and used in the analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Weighted Bag (Traction) | Leg Taping (Taping)
Number analyzed (Participants) | 96 | 95
units on a scale | 5 [0 to 10] | 5 [0 to 10]

3. Secondary Outcome: Time to Foley Expulsion
Description: time from Foley placement until it is spontaneously expulsed from the cervix
Time Frame: an average of 2 hours, up to 12 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Weighted Bag (Traction) | Leg Taping (Taping)
Number analyzed (Participants) | 96 | 95
hours | 1.5 [0.1 to 6.3] | 2.6 [0.2 to 10.8]

4. Other Pre Specified Outcome: Maternal Morbidities
Description: post-partum hemorrhage, clinical chorionamnionitis, endomyometritis, cervical laceration, second procedure, readmission, DVT
Time Frame: 30 days after delivery
Measure: Number; unit: diagnoses
Arm/Group | Weighted Bag (Traction) | Leg Taping (Taping)
Number analyzed (Participants) | 96 | 95
diagnoses | 17 | 16

ADVERSE EVENTS:
Arm/Group | Weighted Bag (Traction) | Leg Taping (Taping)
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/95
Other Adverse Events (participants affected / at risk) | 0/96 | 0/95

LIMITATIONS AND CAVEATS:
Nine patients had minor protocol violations yet were included in the intention to treat analysis. Patients and providers were not be blinded. Our inner city, minority population at a single site may also limit the generalizability of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No